CLINICAL TRIAL: NCT00718822
Title: Does Reduced Oxygen Tension in Embryo Culture Influence Clinical Outcome of ICSI Cycles? A Prospective Randomized Trial
Brief Title: Outcome of Embryo Culture at Two Oxygen Tensions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Maribor (Other)
Collaborators: Slovenian Research Agency (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P3-0327
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2008-07-21 (Estimated); Status verified 2008-07

CONDITIONS: Embryo Development
Keywords: clinical outcome; ICSI cycles; low oxygen; poor responders; pregnancy rate; prospective randomized study

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): 5% oxygen concentration in the culture atmosphere
  Interventions: Other: oxygen concentration in the culture atmosphere
- II (Experimental): 20% oxygen concentration in the culture atmosphere
  Interventions: Other: oxygen concentration in the culture atmosphere

INTERVENTIONS:
Other: oxygen concentration in the culture atmosphere

SUMMARY:
The purpose of this study is to assess whether reduced oxygen tension in embryo culture has any effect on clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* stimulated Intra Cytoplasmic Sperm Injection (ICSI) cycle

Exclusion Criteria:

* less than one mature (metaphase II) oocyte at the time of denudation

Ages: 22 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 647 (Actual)
Dates: Start 2006-08; Primary Completion 2007-06 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate per cycle | 10-11 weeks after embryo transfer

SECONDARY OUTCOMES:
clinical pregnancy rate, implantation rate, early pregnancy loss, fertilization rate, embryo quality

CONTACTS AND LOCATIONS:
Overall Officials: Veljko Vlaisavljević, Prof., Study Chair — University Medical Centre Maribor
Locations (1):
- University Clinical Centre Maribor, Maribor, Slovenia